CLINICAL TRIAL: NCT05902221
Title: Impact of Rifampicin in Treatment Outcome of Cutibacterium Acnes Prosthetic Joint Infections
Acronym: RIFACute
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-APN-02
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Infections Joint Prosthetic
MeSH Terms: interventions — Amoxicillin; Moxifloxacin; Rifampin

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized two-arm (parallel) comparative open-label cohort clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic treatment backbone alone (Active Comparator): Amoxicillin or moxifloxacin to the investigator's discretion
  Interventions: Drug: amoxicillin or moxifloxacin
- Antibiotic treatment backbone + rifampicin (Experimental): Amoxicillin or moxifloxacin to the investigator's discretion + RIMACTAN
  Interventions: Drug: amoxicillin or moxifloxacin + rifampicin

INTERVENTIONS:
Drug: amoxicillin or moxifloxacin — Antibiotic treatment back bone during 12 weeks
  Arms: Antibiotic treatment backbone alone
Drug: amoxicillin or moxifloxacin + rifampicin — Antibiotic treatment back bone during 12 weeks + rifampicin
  Arms: Antibiotic treatment backbone + rifampicin

SUMMARY:
Cutibacterium acnes is involved in nearly 40% of shoulder prosthetic joint infections (PJI). After shoulder prothesis, C. acnes mainly affects hip prosthesis. One recent work from the Lyon (France) bone and joint infections reference center with data focusing mainly on hip and knee PJI has reported that C. acnes is the leading cause of late-onset PJI after coagulase negative staphylococci (CNS) (late acute PJI not considered).

In such late-onset device-related infection, biofilm, as produced by C. acnes during PJI represents a major hurdle on the path to patient's cure. Because biofilm-associated bacteria have a slower metabolism and a lower multiplication rate than planktonic bacteria, antibiotic susceptibility can be hampered.

Rifampicin is an antibiotic with low minimal bactericidal concentration against S. aureus and CNS biofilm-associated bacteria8 which significantly influence patient's outcome during staphylococci PJI.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or =18 years old;
* Monomicrobial, rifampicin susceptible Cutibacterium acnes late total knee arthroplasty (TKA) or hip arthroplasty (total, THA or hemiarthroplasty, HH) or shoulder arthroplasty (total, TSA or hemiarthroplasty, SH) infection treated surgically with single-stage or two-stage revision;
* Isolation of C. acnes on two distinct per-operative samples collected during the single-stage or the two-stage revision
* Based on the antimicrobial susceptibility test of the C. acnes and the medical history of the patient, the PJI can be treated with amoxicillin or moxifloxacin;
* Women considered of childbearing potential (WOCBP) requires use of a highly effective contraceptive measure as intrauterine device (IUD), intrauterine hormone-releasing system (IUS), documented bilateral tubal occlusion, documented vasectomised partner, sexual abstinence. Contraception should be maintained during treatment and until the end of relevant systemic exposure.

Exclusion Criteria:

* Contraindication to Rifampicin (included ongoing treatment contraindicated with rifampicin)
* Contraindication to Amoxicillin AND moxifloxacin (included ongoing treatment contraindicated with these medicines)
* Empirical antibiotic treatment not administered during the 24 hours following revision surgery;
* Inactive empirical antibiotic treatment following surgery according to the AST of the bacteria;
* disease-modifying treatment incompatible with the inducer effect of rifampicin
* Liver cirrhosis;
* Pregnancy: a pregnancy blood test will be performed on all women of childbearing age. The results will be sent to the patient by the doctor of their choice;
* Porphyria;
* Renal insufficiency with GFR < 30ml/min/1.73 m2 (CKD-EPI);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of C. acnes prosthetic joint infections management failure | 24 months after the end of antibiotic treatment
  Defined by Relapse, New infection, early failure
Rate of adverse event linked to rifampicin | during rifampicin treatment
  adverse events will be described by frequency and grade, throughout the treatment (classified according to the CTCAE 5.0.)

SECONDARY OUTCOMES:
Rate of C. acnes prosthetic joint infections probable failure | 24 months after the end of antibiotic treatment
  prosthetic joint infections probable failure suspected in case of specific clinical signs (fistula) and/or inflammatory synovial fluid without microbiological positive results and/or histopathological results after revision without microbiological positive results
Rate of C. acnes prosthetic joint infections management failure | 24 months after the end of antibiotic treatment
  Defined by Relapse, New infection, early failure
Rate of C. acnes prosthetic joint infections management failure | 12 months after the end of antibiotic treatment
  Defined by Relapse, New infection, early failure

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CH Annecy Genevois, Annecy
  - CHU de BORDEAUX, Bordeaux
  - HCL, Lyon
  - AP-HM, Marseille
  - CHU de MONTPELLIER, Montpellier
  - CHU de Nantes, Nantes
  - CHU de NICE, Nice
  - Dianonesses croix saint simon, Paris
  - CHU de Rennes, Rennes
  - CHU Toulouse, Toulouse
  - Ch Tourcoing, Tourcoing
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No
Not planned